CLINICAL TRIAL: NCT00200590
Title: Analgesic Strategies in Newborns Receiving Prostaglandin Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: More important number of SAE in one arms
Sponsor: Nantes University Hospital (Other)
Responsible Party: Dr Véronique Gournay, CHU de Nantes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/03/7-D
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Pain
Keywords: prostaglandin; analgesia; congenital; heart; defect; induced
MeSH Terms: conditions — Pain; Agnosia | interventions — Acetaminophen; Nalbuphine; Morphine

INTERVENTIONS:
Drug: acetaminophen and nalbuphine
Drug: acetaminophen and morphine
Drug: acetaminophen and reduced dosage of prostaglandin

SUMMARY:
This is a randomised trial comparing the efficacy of 3 different analgesic strategies in newborns on prostaglandin for ductus dependent congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Full-term newborn
* Under one month of age
* With ductus dependent congenital heart disease requiring prostaglandin infusion and elevated pain score

Exclusion Criteria:

* Contraindication to either morphine, acetaminophen, or nalbuphine
* Other painful condition
* Poor neurological condition
* Cardiac instability requiring urgent surgery

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2003-12; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Pain score | before inclusion and at 8 hours (H8), H24, H48, H72

SECONDARY OUTCOMES:
Incidence of apnea
Need for mechanical ventilation
Incidence of fever
Pattern of feeding (oral, nasogastric [NG] tubing, parenteral nutrition)

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Gournay, MD, Principal Investigator — Nantes UH
Locations (1):
- Nantes University Hospital, Nantes, France